CLINICAL TRIAL: NCT05165589
Title: Pilot & Exploratory - Validation of Active-Insights Device to Measure Crying Time
Brief Title: Validation of Active-Insights Device to Measure Crying Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioGaia AB (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); ActivInsights (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CSUB0201
Record Dates: First submitted 2021-10-15; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Infant Behavior
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Intervention Model Description: Part 1: 3 subjects for 4 days included to collect initial data for algoritm development for device feasibility evaluation Part 2: 10 subjects for 7 days included to evaluate device feasibility
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Initial data collection for device feasibility (Experimental): 3 subjects for 4 days included to collect initial data for algoritm development for device feasibility
  Interventions: Device: ActiveInsights accelerometer device
- Part 2: Device feasibility (Experimental): 10 subjects for 7 days included to evaluate device feasibility
  Interventions: Device: ActiveInsights accelerometer device

INTERVENTIONS:
Device: ActiveInsights accelerometer device — Accelerometer device

SUMMARY:
To assess the ability of a machine learning algorithm to accurately detect fussing and crying time in infants using accelerometery data collected from a wearable device, compared to the Barr's parent-/caregiver-completed behaviour diary.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 4-12 weeks at screening.
2. Gestational age 37 weeks - 41 weeks at birth.
3. Birth weight appropriate for gestational age (AGA - weight between 10th and 90th percentile) or Large for Gestational Age (LGA - weight above the 90th percentile) determined using WHO Weight-for Age percentile guides.
4. Infant has excessive crying, defined as 3 or more hours per day, during 3 or more days in the preceding week.
5. No birth trauma and nonsyndromic.
6. Readiness and the opportunity for parents/caregivers to fill out a study diary, questionnaires and for infant to wear device.
7. Parent/caregiver with ability to understand and comply with the requirements of the study, as judged by the Investigator.
8. Parent/caregiver willing and able to give informed consent for their and their infant's participation in the study.
9. Infant is considered healthy, following physical exam.

Exclusion Criteria:

1. Infants with failure to thrive, intrauterine growth retardation, haematochezia (blood in the stools), diarrhoea (watery stools that takes the shape of a container > 12x in breastfed and >5 in partially breastfed infants daily), or fever (38.0 degrees).
2. Premature infants (<35 weeks gestation at birth).
3. Infants with congenital heart disease, immunodeficiency, asplenia, cancer, cystic fibrosis, formula-fed infants, and those with liver disease.

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Device feasibility: Comparison of device-generated versus diary-reported crying and fussing time data | 4 days
  Part 1: Comparison of daily crying and fussing time data generated by accelerometer and machine-learning versus crying and fussing time data reported by parental Barrs diary
Device feasibility: Comparison of device-generated versus diary-reported crying and fussing time data | 7 days
  Part 2: Comparison of daily crying and fussing time data generated by accelerometer and machine-learning versus crying and fussing time data reported by parental Barrs diary

SECONDARY OUTCOMES:
Device feasibility: Comparison of device-generated versus diary-reported crying time data | 7 days
  Part 2: Comparison of daily crying time data generated by accelerometer and machine-learning versus crying time data reported by parental Barrs diary
Device feasibility: Comparison of device-generated versus diary-reported fussing time data | 7 days
  Part 2: Comparison of daily fussing time data generated by accelerometer and machine-learning versus fussing time data reported by parental Barrs diary
Device feasibility: Comparison of device-generated versus diary-reported sleeping time data | 7 days
  Part 2: Comparison of daily sleeping time data generated by accelerometer and machine-learning versus sleeping time data reported by parental Barrs diary

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No